CLINICAL TRIAL: NCT02718456
Title: Overcoming Barriers to HIV/AIDS Care and ART Initiation
Acronym: LINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Brandon Guthrie, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000059
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Engagement in HIV Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of care (No Intervention): Standard HIV counseling and referral to care
- CD4 testing (Experimental): Standard HIV counseling and testing plus blood drawn for CD4 testing at time of HIV diagnosis. CD4 results are reported to participants via telephone within 1 week.
  Interventions: Behavioral: Expedited CD4 testing
- CD4 testing plus peer counseling (Experimental): Standard HIV counseling and testing plus blood drawn for CD4 testing at time of HIV diagnosis. CD4 results are reported to participants via telephone within 1 week. Additionally, a trained peer counselor provides supplemental counseling at the time of diagnosis and at the 1 week telephone follow-up.
  Interventions: Behavioral: Expedited CD4 testing; Behavioral: Supplemental peer counseling

INTERVENTIONS:
Behavioral: Expedited CD4 testing
  Arms: CD4 testing; CD4 testing plus peer counseling
Behavioral: Supplemental peer counseling
  Arms: CD4 testing plus peer counseling

SUMMARY:
The study will evaluate interventions to improve engagement in HIV care following HIV diagnosis through a voluntary counseling and testing program. The specific aims are to (1) determine if a VCT-based intervention of CD4 count testing, alone or in combination with peer counseling, improves linkage to HIV/AIDS care; (2) assess the impact of the intervention on ART initiation. The study will recruit 450 HIV-positive individuals from VCTs and randomize a third to standard counseling and referral, a third to receive CD4 testing at the VCT with results return by phone after 1 weeks, and a third to receive the same CD4 testing combined with peer counseling. These combined investigations will create a comprehensive understanding of obstacles to appropriate HIV/AIDS care and result in new interventions to achieve measurable outcomes in applied settings.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older and
* Testing HIV-positive for the first time at a voluntary counseling and testing (VCT) center.
* Willing to receive counseling to encourage linkage to care at a comprehensive care center (CCC).
* Willing to have a CD4 count test conducted at the enrollment visit.
* Willing to have a telephone follow-up where they may receive additional counseling and/or have their CD4 count results returned to them.
* Willing to be contacted over 1 year to determine if they linked to care.

Exclusion Criteria:

* Previous positive HIV test.
* Currently taking antiretroviral medications.
* Currently pregnant (females only).
* Currently participating in another research study or trial.
* Not planning to remain in Nairobi for the next 12 months (not including short trips out of Nairobi).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Number of days from study enrollment until first visit to a comprehensive care center for HIV care. | 1 year
  An interviewer administered questionnaire will be used to determine if each participant visited a comprehensive care center. Is so, the date of the first visit will be recorded. From this, the time from enrollment until first visit to a comprehensive care center will be calculated.
Number of days from study enrollment until initiation of antiretroviral therapy. | 1 year
  An interviewer administered questionnaire will be used to determine if each participant started antiretroviral therapy. Is so, the date of treatment initiation will be recorded. From this, the time from enrollment until treatment initiation will be calculated.

SECONDARY OUTCOMES:
Interviewer-administered questionnaire to determine the number of visits made to a comprehensive care center for HIV care. | 1 year
  Measurement of the number of visits to a comprehensive care center will be made questionnaire administered in an in-person interview at 12 months after enrollment. The total number of visits will be recorded.
Measurement of CD4+ T-cell count. | 1 year
  Each participant's CD4 count will be measure at 1 year after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon L Guthrie, PhD, Principal Investigator — University of Washington
Locations (1):
- Karen Health Center, Nairobi, Kenya